CLINICAL TRIAL: NCT03120533
Title: Therapeutic Iontophoresis of Treprostinil in Systemic Sclerosis Digital UlcErations. A Proof of Concept Study
Brief Title: Treprostinil Iontophoresis in Systemic Sclerosis Digital UlcErations. A Proof of Concept Study
Acronym: TISSUE-PoC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Linksium (Unknown); University Grenoble Alps (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 38RC16.005
Record Dates: First submitted 2017-03-23; First posted 2017-04-19 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Scleroderma, Systemic
Keywords: iontophoresis; treprostinil
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treprostinil (Experimental): the participant will receive 10 days of iontophoresis of treprostinil on a first site, each day the same site.
  Interventions: Drug: Iontophoresis of treprostinil
- Placebo (Placebo Comparator): the participant will receive 10 days of iontophoresis of NaCl on a second site, but the same time than treprostinil
  Interventions: Drug: Iontophoresis of placebo

INTERVENTIONS:
Drug: Iontophoresis of treprostinil — the participant will receive 10 days of iontophoresis of treprostinil on a first site
  Arms: Treprostinil
Drug: Iontophoresis of placebo — the participant will receive 10 days of iontophoresis of NaCl on a second site, but the same time than treprostinil; it's like a design of cross-over study
  Arms: Placebo

SUMMARY:
The study is conducted to confirm the good tolerance of a continuous cathodal iontophoresis of the treprostinil hydrogel administered during 10 days on the pulp of the finger of healthy volunteer and on the ischemic digital ulcerations of Systemic Sclerosis patients, particularly to estimate the cutaneous tolerance of the procedure and the effect on the blood pressure.

DETAILED DESCRIPTION:
Systemic Sclerosis is a rare disease characterized by microvascular affection and cutaneous fibrosis. The digital ulcers are a severe and very invalidating complication. The vascular dysfunction is a key element in the pathogenesis of this disease, preceding the fibrosis. The physiopathology involves a vascular ischemia and mechanical factors or cutaneous calcinoses, or local trauma. The treatment of the digital ulcerations of the Systemic Sclerosis is at first preventive within the a good cutaneous and ungual hygiene, with recourse, as a preventive measure, to Bosentan, an endothelin antagonist. Iloprost by intravenous route is the recommended curative treatment, but patients present very frequent and dose - limiting side effects (headaches, vasomotor flushing, nausea, vomiting, maxillary pains, myalgia).

The paradox is that the decrease of the capillary density and the lower microvascular reactivity limits the distribution of the drug at its site of action when it is administered by intravenous route. High doses are then necessary to reach a sufficient concentration in the region of the wound, which generates side effects. The local administration of the drug could allow to by-pass this problem.

The investigator uses a technique for the topical administration of a vasodilator close to iloprost, treprostinil. This technique is iontophoresis. In the previous clinical trials INFLUX-IT and TIPPS, the investigator showed that the local cutaneous administration of treprostinil by cathodal iontophoresis at 0.03 milliAmper(mA)/cm2 is well tolerated (no local or systematic side effect in healthy volunteer, Systemic Sclerosis patients and diabetics). Iontophoresis induced a steady increase of the cutaneous blood flow of fingers. The investigator also showed that treprostinil was detectable in the dermis until 8 hours after the iontophoresis, without significant increase in the plasma. Thus, daily repeated iontophoresis on 10 days on ulcerated areas could allow to obtain therapeutic tissular concentrations.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

* Age of at least 18 years
* Existence of a contraceptive method for women of child-bearing age
* Person affiliated to social security or beneficiary of such a scheme
* Signed consent form

Systemic sclerosis patients:

* Systemic sclerosis meeting the EULAR criteria.
* Presence of 1 ischemic digital cutaneous ulceration , with digital ulcer classified as "active ulcers" according to the North American working group definition: epithelial denudation is clearly Visible at one place and the bed of de-epithelialized ulcer can be seen; Ulcerations distal to the proximal interphalangeal joint, not associated with calcinosis or bony relief.
* Ulcers whose major axis measured with the electronic caliper is ≥ 2 mm
* Age greater than or equal to 18 years
* Existence of a contraceptive method for women of reproductive age
* A person who is or is a beneficiary of social security
* Informed and signed consent signed by the patient or his / her legal representative.

Exclusion Criteria:

Healthy Volunteers

* Treprostinil contraindications: Known hypersensitivity to treprostinil or any of the excipients, Pulmonary arterial hypertension related to veno-occlusive disease, Congestive heart failure due to severe left ventricular dysfunction, Severe hepatic insufficiency (Child-Pugh stage C), Evolving gastrointestinal ulcer, intracranial hemorrhage, recent trauma or other clinical condition that may lead to bleeding, Congenital or acquired valvular abnormalities with cardiac repercussions, Severe ischemic heart disease or unstable angina; Myocardial infarction in the last six months; Decompensated cardiac insufficiency not medically controlled; Severe arrhythmias; Cerebrovascular lesions (such as transient ischemic attack, stroke) that occurred within the last three months.
* Persons referred to in Articles L1121-5 to L1121-8 of the French Public health Code: pregnant woman, parturient, nursing mother, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure, can not Be included in clinical trials.
* Subject in an exclusion period from another study,
* Subject who would receive more than 4500 euros of compensation due to his participation in other biomedical research in the 12 months preceding this study

Systemic sclerosis patients:

* Iloprost cure carried out in the previous month or planned in the following month.
* Initiation or change of dosage of bosentan, sildenafil or calcium channel blockers in the previous month or in the following month
* Digital Sympathectomy or botulinum toxin injection planned in the following month.
* Clinically superinfected digital ulcers
* Treprostinil contraindications: Known hypersensitivity to treprostinil or any of the excipients, Pulmonary arterial hypertension related to veno-occlusive disease, Congestive heart failure due to severe left ventricular dysfunction, Severe hepatic insufficiency (Child-Pugh stage C), Evolving gastrointestinal ulcer, intracranial hemorrhage, recent trauma or other clinical condition that may lead to bleeding, Congenital or acquired valvular abnormalities with cardiac repercussions, Severe ischemic heart disease or unstable angina; Myocardial infarction in the last six months; Decompensated cardiac insufficiency not medically controlled; Severe arrhythmias; Cerebrovascular lesions (such as transient ischemic attack, stroke) that occurred within the last three months.
* Persons referred to in Articles L1121-5 to L1121-8 of the French Public health Code: pregnant woman, parturient, nursing mother, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure, can not Be included in clinical trials.
* Subject in an exclusion period from another study,
* Subject who would receive more than 4500 euros of compensation due to his participation in other biomedical research in the 12 months preceding this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Number of side-effects graduated according to NIH CTCAE 4.03 | every day of iontophoresis from day 0 to day 9
  Side effects will be reported according to NIH CTCAE 4.03, particularly " Skin and subcutaneous tissue disorders " et " Vascular disorders ".

SECONDARY OUTCOMES:
Pharmacodynamical effect of iontophoresis of treprostinil hydrogel in healthy volunteers on pulp finger, leg and foot | day 0
  area under curve of the increase of the flow after the iontophoresis of the gel of treprostinil compared to the iontophoresis of Sodium Chloride (NaCl) measured by laser speckle imaging
Pharmacodynamical effect of 10 days of iontophoresis of treprostinil hydrogel in systemic sclerosis patients | day 0 and day 9
  cutaneous vascular conductance after the iontophoresis of the gel of treprostinil compared to the iontophoresis of NaCl measured by laser speckle imaging
Pharmacodynamical effect of 10 days of iontophoresis of treprostinil hydrogel in systemic sclerosis patients | day 0 and day 9
  Area under curve of the cutaneous flow after the iontophoresis of the gel of treprostinil compared to the iontophoresis of NaCl measured by laser speckle imaging
Effect of iontophoresis of treprostinil hydrogel on peri and intra ulcer flow | day 0 and day 9
  cutaneous vascular conductance of the ulceration areas after the iontophoresis of the gel of treprostinil compared to the iontophoresis of NaCl measured by laser speckle imaging
Systemic diffusion of the treprostinil hydrogel administered by iontophoresis | day 0 and day 9
  Plasmatic concentration of treprostinil

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc CRACOWSKI, MD,PhD, Principal Investigator — CIC 1406
Locations (1):
- Grenoble Alps University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaillard-Bigot F, Roustit M, Blaise S, Cracowski C, Seinturier C, Imbert B, Carpentier P, Cracowski JL. Treprostinil Iontophoresis Improves Digital Blood Flow during Local Cooling in Systemic Sclerosis. Microcirculation. 2016 Apr;23(3):266-70. doi: 10.1111/micc.12272. PMID 26833587
- [Background] Hellmann M, Roustit M, Gaillard-Bigot F, Cracowski JL. Cutaneous iontophoresis of treprostinil, a prostacyclin analog, increases microvascular blood flux in diabetic malleolus area. Eur J Pharmacol. 2015 Jul 5;758:123-8. doi: 10.1016/j.ejphar.2015.03.066. Epub 2015 Apr 3. PMID 25843412
- [Background] Kotzki S, Roustit M, Arnaud C, Godin-Ribuot D, Cracowski JL. Effect of continuous vs pulsed iontophoresis of treprostinil on skin blood flow. Eur J Pharm Sci. 2015 May 25;72:21-6. doi: 10.1016/j.ejps.2015.02.012. Epub 2015 Feb 21. PMID 25712367
- [Background] Roustit M, Gaillard-Bigot F, Blaise S, Stanke-Labesque F, Cracowski C, Seinturier C, Jourdil JF, Imbert B, Carpentier PH, Cracowski JL. Cutaneous iontophoresis of treprostinil in systemic sclerosis: a proof-of-concept study. Clin Pharmacol Ther. 2014 Apr;95(4):439-45. doi: 10.1038/clpt.2013.255. Epub 2014 Jan 23. PMID 24458011
- [Background] Kotzki S, Roustit M, Arnaud C, Boutonnat J, Blaise S, Godin-Ribuot D, Cracowski JL. Anodal iontophoresis of a soluble guanylate cyclase stimulator induces a sustained increase in skin blood flow in rats. J Pharmacol Exp Ther. 2013 Sep;346(3):424-31. doi: 10.1124/jpet.113.205484. Epub 2013 Jul 9. PMID 23838678
- [Background] Blaise S, Roustit M, Hellmann M, Millet C, Cracowski JL. Cathodal iontophoresis of treprostinil induces a sustained increase in cutaneous blood flux in healthy volunteers. J Clin Pharmacol. 2013 Jan;53(1):58-66. doi: 10.1177/0091270011434352. Epub 2013 Jan 24. PMID 23400744
- [Background] Blaise S, Roustit M, Millet C, Ribuot C, Boutonnat J, Cracowski JL. Cathodal iontophoresis of treprostinil and iloprost induces a sustained increase in cutaneous flux in rats. Br J Pharmacol. 2011 Feb;162(3):557-65. doi: 10.1111/j.1476-5381.2010.01045.x. PMID 20860718